CLINICAL TRIAL: NCT03954756
Title: Phase II Clinical Study of the Combination of Apatinib and PD1 in Treating Advanced Gastric Cancer
Brief Title: Exploratory Clinical Study of Apatinib and PD-1 in Treating Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APD-L0315
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib and PD-1 (Experimental): Every patients will received apatinib orally every day and PD-1 200mg (3mg/kg for underweight patients) iv every 2 weeks until disease progression or intolerance of side effect
  Interventions: Drug: Apatinib and PD1

INTERVENTIONS:
Drug: Apatinib and PD1 — 1. Apatinib starting dose of 500mg, qd, oral, taken half an hour after a meal
  2. PD-1 was administered 200mg (3mg/kg for underweight patients) iv every 2 weeks.

SUMMARY:
The Purpose of This Study is to Evaluate the Efficacy and Safety of Apafitini Combined With PD1 in Patients With Advanced Gastric Cancer After Second-line Treatment Failure, Thus Providing More Options for Patients With Advanced Gastric Cancer.

DETAILED DESCRIPTION:
Patients will received apatinib orally every day and PD-1 200mg (3mg/kg for underweight patients) iv every 2 weeks. The efficacy and safety will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients join the study voluntarily, sign a consent form, have good compliance, and comply with follow-up.
2. To be confirmed to meet the clinical diagnosis standard, histologically or cytologically confirmed advanced Gastric Cancer.
3. Failure of the second-line standard treatment regimen (disease progression), >14 days from the last chemotherapy, chemotherapy regimen including fluorouracil (5-FU / capecitabine / teggio), oxaliplatin and irinotecan; Acceptable or not received bevacizumab/cetuximab/regofenib treatment.
4. Aged 18-70 years old, both genders.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
6. Life expectancy of at least 3 months.
7. Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria.If the lesion receiving local therapy (radiotherapy, radiofrequency, interventional therapy, etc.) is the only lesion, definite imaging progress is required.
8. the main organ functions of the patient shall meet the following standards within 7 days before treatment：Blood routine examination standard (without blood transfusion within 7 days before enrollment）Hemoglobin ≥ 70 g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ PLT）≥80×109/L；Biochemical examination shall meet the following standards:serum total bilirubin (TBIL)≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal(ULN)；Serum creatinine (Cr)≤1.5ULN or creatinine removal rate (CCr)≥60ml/min；
9. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; the serum or urine pregnancy test is negative within 7 days prior to study enrollment and must be Non-lactating patients; males should agree to patients who must use contraception during the study period and within 6 months after the end of the study period。

Exclusion Criteria:

1. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents(within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg；
2. Diabetes blood sugar control is poor；
3. Acute phase of cerebral infarction, or recovery period <2 months；
4. Has a variety of factors that affect the absorption of oral drugs (such as inability to swallow, nausea and vomiting, chronic diarrhea and intestinal obstruction);
5. Patients with a risk of gastrointestinal bleeding may not be enrolled, including the following: (1) active digestive ulcer lesions and fecal occult blood (++); (2) nausea and hematemesis within 2 months Medical history. Simple fecal occult blood (+) is not an exclusion criterion；
6. Coagulation abnormalities （INR>1.5×ULN，APTT>1.5×ULN）,with bleeding tendency;
7. Urine protein ≥ ++ or confirmed 24 hour urine protein quantitation > 1.0 g；
8. Pregnant or lactating women;
9. Within 2 weeks after treatment with cytotoxic drugs and radiotherapy;Has taken two or more oral targeted drugs；
10. Except for other malignant tumors, basal cell carcinoma of the skin and cervical cancer in situ in the past 5 years；
11. The investigator believes that there are any conditions that may damage the subject or result in the subject being unable to meet or perform the research request；
12. Patients with severe liver and kidney dysfunction (grade 4) should be excluded;
13. Those who are allergic to any component of apafitini mesylate should be excluded;
14. Mental disorders history, or psychotropic drug abuse history；
15. Previous use of regorafenib is not an exclusion criterion；
16. According to the investigator's judgment, there are people with concomitant diseases that seriously endanger the safety of the patient or affect the patient's completion of the study;
17. Surgery was performed within 4 weeks prior to the start of treatment, or patients with major trauma or fractures. Or there is an unhealed wound before treatment;
18. Patients with severe heart disease, such as grade III or above (NYHA standard) congestive heart failure, or grade III or above (CCS standard) angina, or a history of myocardial infarction within 6 months prior to treatment, or an arrhythmia requiring medication;
19. The patient has brain metastasis, meningeal metastasis;
20. Active HBV infection and rejection of formal antiviral therapy;
21. Active tuberculosis;
22. Participants who have participated in any drug or medical device clinical trial within 1 month prior to the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | up to 2 year

SECONDARY OUTCOMES:
Objective response rate | up to 2 year
  Defined as the proportion of patients with a documented complete response, and partial response (CR
  + PR
Disease control rate | up to 2 year
  The time from the start of randomization to the first tumor recurrence/metastasis or the death of the subject for any reason
Overall survival | up to 2 year
  From date of randomization until the date of death from any cause